CLINICAL TRIAL: NCT02067923
Title: ITN0127AI Autoimmunity-blocking Antibody for Tolerance in Recently Diagnosed Type 1 Diabetes (AbATE) Follow-Up Study
Brief Title: AbATE Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1310012954
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1D; type 1 diabetes; type 1 diabetes mellitus; juvenile diabetes; autoimmune diabetes; autoimmune; anti-CD3 mAb; mAb hOKT3g1(Ala-Ala); teplizumab
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anti-CD3 mAb Plus Diabetes Standard of Care Group: This group of individuals received treatment in the original AbATE study.
- Diabetes Standard of Care Group: During the original AbATE study these individuals received standard care.

SUMMARY:
This study proposes to conduct a non-interventional, multi-center trial that will look at C-peptide results from one or two Mixed Meal Tolerance Tests (MMTT) in participants who received anti-CD3 treatment or placebo on the Abate ITN027AI trial. Anti-CD3 monoclonal antibody is a humanized antibody that is commonly used to prevent organ rejection. It was give in order to determine whether anti-CD3 mAb treatment can halt the progression of newly diagnosed type 1 diabetes.

The overall hypothesis of this study is there will be less change in c-peptide levels of the previously treated group versus the control group.

DETAILED DESCRIPTION:
We propose to conduct a non-interventional multi-center trial that will look at C-peptide results from one or two Mixed Meal Tolerance Tests (MMTT) in participants who received anti-CD3 treatment or placebo on the Abate ITN027AI trial. The first few subjects went on the trial late in 2005 and the last subjects were enrolled in 2009.The mixed meal tolerance tests will coincide with approximately 4 years and 6 years post ITN027AI study completion for each participant. Those participants, who completed the ITN027AI study in 2007 and 2008, will only have a single MMTT.

We plan to enroll approximately 77 subjects at 5 sites who were previously active with ITN027AI.. Both the drug treated and the control group participants will be invited to participate. Along with Yale University these sites include, the University of California-San Francisco, University of Colorado-Barbara Davis, Benaroya Research Institute, and Pacific Northwest Research Institute -University of Washington. The investigators of each of these sites will be asked to contact their patients who were originally on the ITN027AI study.

Subjects will be contacted via email or phone to see if they would be interested in participating on this Abate follow-up study. Eligible participants will come to the Yale University Church St. Research Unit or other participating ITN study site for either 1 or 2 mixed meal tolerance tests to determine their current c-peptide status. The available sites for participants to go to include: Yale University, University of California-San Francisco, University of Colorado-Barbara Davis Center, Benaroya Research Institute and Pacific Northwest-University of Washington.

This first visit will consist of the following: an explanation of the study, an assessment of inclusion/exclusion criteria and documentation of informed consent. If the subject meets the inclusion/exclusion criteria, a complete medical history will be obtained, physical examination including vital signs, urine pregnancy test if a female of childbearing potential and an assessment of concomitant medications. The subject will then have a Mixed Meal Tolerance Tests (MMTT) with a possible 2nd MMTT with C-Peptide and glucose measurements a year later based on how long it has been since they were on the ITN027AI Study.The subject will also have a 4 hour urine collection for C-peptide and creatinine during this MMTT. If a repeat MMTT is done a year later then another 4 hour urine sample during the MMTT will be collected for C-peptide and Creatinine measurement.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation on either the treatment or the control arm of the Abate ITN027AI trial
* Signed Informed Consent

Exclusion Criteria:

* Inability or unwillingness to give informed consent
* Participation in an investigational treatment trial within the last 6 weeks before enrollment
* Ongoing major systemic illness.
* Clinically active serious infections.
* Any medical condition that in the opinion of the investigator would interfere with safe completion of the trial.
* Positive pregnancy test in menstruating women
* Actively breast feeding

Ages: 10 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The investigators will contact their patients who were originally on the ITN027AI (AbATE) study. Subjects will be contacted via email or phone to see if they would be interested in participating on this Abate follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
Mixed Meal Tolerance Test (MMTT) C-peptide levels | 1 Study Day
  Labs will be obtained to assess beta cell function via c-peptide levels and glucose at 11 time points during the mixed meal tolerance test. Blood samples will be obtained prior to the start of the mixed meal tolerance test to assess auto-antibody status and HbA1c. Approximately 60 cc's of blood will also be obtained for PBMC's and future studies as related to the immunology and genetics of T1DM. A 4 hour urine sample during the MMTT will be collected for C-peptide and Creatinine measurement. We plan to determine the relationship between this measurement and the insulin secretory response.

SECONDARY OUTCOMES:
Safety experience | 1 Study Day
  To determine the safety experience and diabetes specific clinical parameters in previous participants in the ITN027 trial via the history of hospitalizations and other adverse events since the participants came of the original ITN027AI Treatment Trial.

CONTACTS AND LOCATIONS:
Overall Officials: Kevan Herold, MD, Principal Investigator — Yale University
Locations (1):
- Church Street Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Perdigoto AL, Preston-Hurlburt P, Clark P, Long SA, Linsley PS, Harris KM, Gitelman SE, Greenbaum CJ, Gottlieb PA, Hagopian W, Woodwyk A, Dziura J, Herold KC; Immune Tolerance Network. Treatment of type 1 diabetes with teplizumab: clinical and immunological follow-up after 7 years from diagnosis. Diabetologia. 2019 Apr;62(4):655-664. doi: 10.1007/s00125-018-4786-9. Epub 2018 Dec 19. PMID 30569273